CLINICAL TRIAL: NCT00006487
Title: A Phase I Study Of Tirapazamine/Cisplatin/Etoposide And Concurrent Thoracic Radiotherapy For Limited Stage Small Cell Lung Cancer
Brief Title: S0004: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Limited-stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068318; U10CA032102 (NIH); S0004 (Other: SWOG)
Record Dates: First submitted 2000-11-06; First posted 2004-04-02 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Tirapazamine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemo/RT with tirapazamine (Active Comparator): induction and consolidation: cisplatin, etoposide, tirapazamine, radiation therapy
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: tirapazamine; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — During induction: 50 mg/m2/day, IV on Days 1, 8, 29, 36. 1 hour infusion
  During consolidation: 60 mg/m2, IV on Day 1 only at approximately Week 11, Week 14. 1 hour infusion.
  Other Names: platinol
Drug: etoposide — During induction: 50 mg/m2/day, IV on Days 1 - 5, 29 - 33. 1 hour infusion
  During consolidation: 120 mg/m2, IV on Days 1, 2 and 3 at approximately Week 11, Week 14. 1 hour infusion.
  Other Names: VP-16
Drug: tirapazamine — During induction:
  Phase I low dose: 260 mg/m2/day, IV on Days 1, 8, 29, 36. 1 hour infusion
  Phase II high dose: 330 mg/m2/day, IV on Days 1, 8, 29, 36 1 hour infusion
  During consolidation:
  330 mg/ m2, IV Day 1 only at approximately Week 11, Week 14. 1 hour infusion.
Radiation: radiation therapy — Radiotherapy should begin within 1 - 3 hours after completion of TPZ infusion on Day 1 of Cycle 1 of induction chemotherapy as outlined above. Computed tomography based treatment planning is strongly recommended.The primary tumor, adjacent mediastinum and other targeted lymph nodes shall receive 4,500 cGy in 25 fractions, five days/week at 180 cGy daily. A 1,600 cGy boost to areas of gross disease will be delivered through reduced off-spinal cord fields in eight fractions, five days/week at 200 cGy daily.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of tirapazamine, cisplatin, and etoposide concurrently with radiotherapy in patients with limited stage small cell lung cancer.
* Determine the toxicities of this treatment regimen in these patients.
* Determine the response rate in these patients treated with this regimen.

OUTLINE: Patients are assigned to one of two induction therapy arms.

* Arm I: Patients receive induction chemotherapy consisting of low-dose tirapazamine IV over 1 hour and cisplatin IV over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Patients also undergo radiotherapy concurrently with chemotherapy 5 consecutive days a week for 7 weeks beginning on day 1.
* Arm II: Patients receive induction chemotherapy consisting of high-dose tirapazamine, cisplatin, etoposide, and radiotherapy as in arm I.

Patients with stable or responding disease then receive consolidation therapy consisting of tirapazamine IV over 1 hour and cisplatin IV over 1 hour on day 1 of weeks 11 and 14 and etoposide IV over 1 hour on days 1-3 of weeks 11 and 14.

Patients are followed every 2 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 50 patients (25 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed limited stage small cell lung cancer (SCLC)
* No malignant pericardial or pleural effusions, including any of the following:

  * Cytologically positive effusions
  * Exudative effusions not attributable to other etiologies
* No brain metastases
* Disease (measurable or non-measurable) must be present outside the area of prior surgical resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than ULN OR
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No symptomatic sensory neuropathy grade 1 or greater
* No other malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other stage I or II cancer in complete remission
* No other medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for SCLC

Chemotherapy:

* No prior systemic chemotherapy for SCLC

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior thoracic radiotherapy for SCLC

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior thoracic or other major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and Toxicity | toxicity is assessed weekly
  If ten or more patients experience either Grade 3 or greater esophagitis or pneumonitis at any dose level, the trial will be stopped. Nine or fewer patients experiencing either of these toxicities will be evidence that the dose can be escalated to the next level.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu X. Le, MD, Study Chair — Stanford University
Locations (87):
- United States (87):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Cancer Center and Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Le QT, McCoy J, Williamson S, Ryu J, Gaspar LE, Edelman MJ, Dakhil SR, Sides SD, Crowley JJ, Gandara DR; Southwest oncology group. Phase I study of tirapazamine plus cisplatin/etoposide and concurrent thoracic radiotherapy in limited-stage small cell lung cancer (S0004): a Southwest Oncology Group study. Clin Cancer Res. 2004 Aug 15;10(16):5418-24. doi: 10.1158/1078-0432.CCR-04-0436. PMID 15328179